CLINICAL TRIAL: NCT00707668
Title: Chung-ju Metabolic Disease Cohort (CMC) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kun-Ho Yoon, Professor, The Catholic University of Korea
Other Study IDs: KCMC07OT076
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Metabolic Diseases
Keywords: Diabetes; metabolic syndrome; dyslipidemia; osteoporosis
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus; Metabolic Syndrome; Dyslipidemias; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Serum Whole blood Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Control: Chung-ju cohort populations aged over 30 year-old

SUMMARY:
This is an observational study on the prevalence and incidence of diabetes and osteoporosis in a rural area of Korea.

DETAILED DESCRIPTION:
Diabetes, metabolic syndrome and dyslipidemia are common and rapidly increasing in Asia. Our group constructed a cohort in Chung-ju city, a rural area in Korea, to observe the prevalence of metabolic diseases and its risk factors since 2003. About 12,000 subjects participated in this cohort study till 2006. Now, we are planning to follow-up these subjects and provide health examinations from May, 2007 to Feb, 2011. The prevalence and incidence of metabolic diseases including diabetes, hypertension, metabolic syndrome, dislipidemia and osteoporosis will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 30 years of age living in Chung-ju city (who participated in 2003-2006 cohort study)

Exclusion Criteria:

* age under 30
* subjects with known diabetes

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 30 years of age living in Chung-ju city
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2007-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of diabetes | 4 years

SECONDARY OUTCOMES:
The prevalence of metabolic syndrome, dyslipidemia and osteoporosis | 4 years
Insulin sensitivity and resistance of Korean subjects | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, M.D., Ph.D., Study Director — Kangnam St.Mary's hospital
Locations (1):
- Chung-ju health care center, Chungju, Chungchungbook-do, South Korea

REFERENCES:
- [Background] Kwon HS, Park YM, Lee HJ, Lee JH, Choi YH, Ko SH, Lee JM, Kim SR, Kang SY, Lee WC, Ahn MS, Noh JH, Kang JM, Kim DS, Yoon KH, Cha BY, Lee KW, Kang SK, Son HY. Prevalence and clinical characteristics of the metabolic syndrome in middle-aged Korean adults. Korean J Intern Med. 2005 Dec;20(4):310-6. doi: 10.3904/kjim.2005.20.4.310. PMID 16491829